CLINICAL TRIAL: NCT02090036
Title: Efficacy and Safety of a Single Low-dose Primaquine Added to Standard Artemether-lumefantrine Treatment for the Clearance of Plasmodium Falciparum Gametocytes.
Brief Title: Efficacy and Safety of a Single Low-dose Primaquine for the Clearance of Gametocytes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Richard Mwaiswelo, Investigator, Muhimbili University of Health and Allied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1.0.2014
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Plasmodium Falciparum
Keywords: Efficacy; Safety; Primaquine; Artemether-lumefantrine; Gametocytes
MeSH Terms: conditions — Malaria, Falciparum | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- artemether-lumefantrine+placebo (Active Comparator): In the artemether-lumefantrine arm, the first dose of artemether-lumefantrine will be administered concomitantly with a single-dose placebo. A volume of normal saline will be measured based on weight bands and then will be given to patients.
  Interventions: Drug: Placebo (For artemether-lumefantrine arm)
- artemether-lumefantrine+primaquine (Experimental): All the recruited patients will be treated with a six doses, 3 days artemether-lumefantrine treatment regimen. However, patients randomized to the artemether-lumefantrine+primaquine arm will be given 0.25 mg/kg single-dose primaquine concomitantly with artemether-lumefantrine first dose.
  Interventions: Drug: Primaquine (For artemether-lumefantrine+primaquine arm)

INTERVENTIONS:
Drug: Primaquine (For artemether-lumefantrine+primaquine arm) — A 0.25 mg/kg single-dose primaquine will be administered concomitantly with the first dose of artemether-lumefantrine in all patients randomized into the artemether-lumefantrine+primaquine arm.
  Arms: artemether-lumefantrine+primaquine
Drug: Placebo (For artemether-lumefantrine arm) — Volume of normal saline mixed with coloured fruit juice measured based on weight bands will be given orally concomitantly with first dose of artemether-lumefantrine.
  Arms: artemether-lumefantrine+placebo

SUMMARY:
The purpose of this study is to assess efficacy and safety of a single low-dose Primaquine added to standard artemether/lumefantrine treatment for the clearance of Plasmodium falciparum gametocytes among patients with uncomplicated malaria aged 1 year and above regardless of their G6PD status.

DETAILED DESCRIPTION:
The current gained successes in malaria control are accredited partly to the availability of efficacious and fast acting artemisinins which are also potent against P. falciparum young gametocytes. Nonetheless, mature gametocytes may persist after treatment, contributing to malaria transmission. Conversely, artemisinin resistance is confirmed in South-east Asia, and it may spread to Africa. New control tools have to be integrated to sustain the gained successes, further reduce transmission and curb the spread of resistance.

Primaquine has strong gametocytocidal effect against mature gametocytes and when added to schizonticidal drugs such as artemether-lumefantrine (AL), it rapidly shorten gametocytes carriage duration, halting disease transmission. Nonetheless, its wide scale use has been hampered by a dose-dependent acute hemolytic anemia it causes in glucose-6-phosphate dehydrogenase (G6PD) deficient individuals. Conversely, Artemisinins potentiate primaquine activities, thus a low dose of primaquine would be able to clear falciparum gametocytes.

The World Health Organization recommends addition of 0.25 mg/kg single-dose primaquine to Artemisinin based combination therapies in malaria endemic areas including Africa without testing for G6PD status. Nonetheless, the recommendation, relies on historical data from South-East Asia and among African Americans in the United States. Therefore, this study plans to assess safety and efficacy of 0.25 mg/kg single-dose primaquine added to a standard AL treatment against P. falciparum gametocytes clearance among patients with uncomplicated malaria aged 1 year and above regardless of their G6PD status..

ELIGIBILITY:
Inclusion Criteria:

* Age of 1 year and above and neither pregnant nor breast feeding.
* Weight over 10 kg.
* Body temperature ≥37.5°C) or history of fever in the last 24 hours.
* P. falciparum mono-infection.

Exclusion Criteria:

* Evidence of severe illness malaria or danger signs.
* Known allergy to study medications.
* Hemoglobin <8 g/dl.
* Antimalarials taken within last 2 weeks.
* Blood transfusion within last 90 days and evidence of recent use (within 14 days)of or will be taking other drugs known to cause hemolysis in G6PD deficient subjects.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of days per treatment arm for gametocytes to become undetectable using Quantitative nucleic acid sequence based assay (QT-NASBA). | 14 days

SECONDARY OUTCOMES:
Mean maximal fall in hemoglobin (g/dl) from enrolment to day 28 of follow-up defined as mean greatest negative difference in hemoglobin per treatment arm. | 28 days.

OTHER OUTCOMES:
Proportion of patients with urine color change score ≥ 5 using Hillmen Urine Colour Chart, per treatment arm. | 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Martensson, PhD, Study Director — Karolinska Institutet
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Mwaiswelo R, Ngasala B, Jovel I, Xu W, Larsson E, Malmberg M, Gil JP, Premji Z, Mmbando BP, Martensson A. Prevalence of and Risk Factors Associated with Polymerase Chain Reaction-Determined Plasmodium falciparum Positivity on Day 3 after Initiation of Artemether-Lumefantrine Treatment for Uncomplicated Malaria in Bagamoyo District, Tanzania. Am J Trop Med Hyg. 2019 May;100(5):1179-1186. doi: 10.4269/ajtmh.18-0729. PMID 30860013
- [Derived] Mwaiswelo R, Ngasala B, Jovel I, Aydin-Schmidt B, Gosling R, Premji Z, Mmbando B, Bjorkman A, Martensson A. Adding a single low-dose of primaquine (0.25 mg/kg) to artemether-lumefantrine did not compromise treatment outcome of uncomplicated Plasmodium falciparum malaria in Tanzania: a randomized, single-blinded clinical trial. Malar J. 2016 Aug 26;15(1):435. doi: 10.1186/s12936-016-1430-3. PMID 27565897
- [Derived] Mwaiswelo R, Ngasala BE, Jovel I, Gosling R, Premji Z, Poirot E, Mmbando BP, Bjorkman A, Martensson A. Safety of a single low-dose of primaquine in addition to standard artemether-lumefantrine regimen for treatment of acute uncomplicated Plasmodium falciparum malaria in Tanzania. Malar J. 2016 Jun 10;15:316. doi: 10.1186/s12936-016-1341-3. PMID 27287612